CLINICAL TRIAL: NCT07108114
Title: A Phase 1 Dose-Escalation Study of SLV-324 in Subjects With Metastatic Solid Tumors
Brief Title: SLV-324 Treatment of Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Solve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLV-324-01Tx
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Solid Tumors
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: In this study, a BOIN design with a target DLT rate for the MTD of 27% and an estimated maximum sample size of ~70 subjects will be used to guide the dose escalation and determine the RDR of SLV-324.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SLV-324 intravenous (IV infusion) (Experimental): SLV-324 will be administered at different dose levels in dose-escalation cohorts and at the RDR in dose expansion cohorts
  Interventions: Drug: SLV-324 intravenous (IV infusion)

INTERVENTIONS:
Drug: SLV-324 intravenous (IV infusion) — SLV-324 will be administered as an IV infusion

SUMMARY:
This is a Phase 1 dose-escalation study evaluating the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and efficacy of SLV-324 across a range of dose levels when administered to subjects with metastatic solid tumors.

DETAILED DESCRIPTION:
A Bayesian optimal interval (BOIN) design with a target dose-limiting toxicity (DLT) rate for the maximum tolerated dose (MTD) of 27% and an estimated maximum sample size of ~70 subjects will be used to guide the dose escalation and determine the recommended dosing regimen (RDR) of SLV-324.

SLV-324 will be administered intravenously (IV) in repeated cycles. Treatment will continue until progressive disease or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women (as appropriate for cancer type) of age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Histologically or cytologically confirmed diagnosis of solid tumor as documented in medical records.
4. Presence of metastatic disease that has progressed during or following previous treatment.
5. Presence of radiographically measurable disease.
6. Prior receipt of commercially available therapies that are indicated for the subject's cancer and have demonstrated survival benefit for that indication.
7. Availability of tumor tissue from a fresh tumor biopsy obtained by a core needle, excisional, or incisional biopsy; or punch biopsy (for cutaneous disease); or archival tumor sample from a previous biopsy.
8. Availability of computed tomography (CT) or magnetic resonance imaging (MRI) of chest, abdomen, and pelvis, and/or fluorodeoxyglucose (FDG) positron emission tomography (PET)/CT (if appropriate for tumor type) (with PET from base of the skull to mid-thigh, if performed) within 35 days before study drug administration.
9. Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥1 week before the start of study drug administration.
10. Adequate hematological profile.
11. Adequate coagulation profile.
12. Adequate hepatic profile.
13. Adequate renal function.
14. Negative viral serology or adequate therapy for human immunodeficiency virus (HIV), hepatitis B (HBV), and hepatitis C (HCV) infection.
15. For female subjects of childbearing potential, a negative serum pregnancy test.
16. For female subjects of childbearing potential, willingness to use a protocol-recommended method of contraception from the start of the screening period until ≥6 months after the final dose of study therapy.
17. For male subjects who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception, willingness to use a protocol-recommended method of contraception from the start of study therapy until ≥6 months after the final dose of study therapy and to refrain from sperm donation from the start of study therapy until ≥12 months after administration of the final dose of study therapy.
18. Willingness and ability of the subject to comply with scheduled visits, the drug administration plan, protocol-specified laboratory tests, other study procedures (including required tumor biopsy/aspirations and/or radiographic studies), and study restrictions.
19. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

1. Malignancy involving the central nervous system unless brain metastases have been previously treated with radiotherapy, have been stable for ≥4 weeks, and do not require corticosteroids.
2. Presence of another cancer with disease manifestations or therapy that could adversely affect subject safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
3. Uncontrolled ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infection) at the time of start of study therapy.
4. Significant cardiovascular event or comorbidity.
5. Significant screening ECG abnormalities.
6. Pregnancy or breastfeeding.
7. Major surgery within 4 weeks before the start of study therapy.
8. Use of a strong inhibitor or inducer of CYP3A4 or CYP1A2.
9. Use of a drug known to prolong the QT interval within 7 days prior to the start of study drug administration.
10. Concurrent participation in another therapeutic or imaging clinical trial.
11. Other conditions likely to interfere with a subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
MTD or RDR | Through the duration of treatment, up to approximately 18 months
  Determination of the MTD (maximum tolerated dose) and/or RDR (recommended dosing regimen) for SLV-324

SECONDARY OUTCOMES:
SLV-324 Administration as Assessed by Prescribing Records | Through the duration of treatment, up to approximately 18 months
  Number of infusions prescribed and administered, body-weight-adjusted and total doses administered, duration of infusions, and number of infusion delays or interruptionsSLV-324 administration as assessed by prescribing records
SLV-324 Safety | Up to approximately 18 months.
  Collection of type, frequency, severity, timing of onset, duration, and relationship to study drug of any treatment-emergent adverse events (TEAEs), laboratory abnormalities, vital sign/oxygen saturation abnormalities, adverse electrocardiogram (ECG) findings, DLTs (dose-limiting toxicities), serious adverse events (SAEs), or adverse events (AEs) leading to interruption, modification, or discontinuation of study drug administration.
Evaluation of use of supportive care and other concomitant medications | Through the duration of treatment, up to approximately 18 months
  Type, frequency, and timing of use of supportive care and other concomitant medications
SLV-324 Pharmacokinetics: Maximum Concentration (Cmax) | Varying timepoints through the duration of treatment, up to approximately 18 months
  Cmax of SLV-324 antibody-drug conjugate, total antibody, and free payload
Immunogenicity | Varying timepoints through the duration of treatment, up to approximately 18 months
  Measurement of changes in titers of circulating SLV-324-reactive antibodies (as assessed using immunoassay methods)
Objective Response Rate (ORR) | Through the duration of treatment, up to approximately 18 months
  ORR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR).
Time to Response (TTR) | Up to approximately 36 months
  TTR: interval from the start of study drug administration to the first documentation of objective tumor regression.
Duration of Response (DOR) | Up to approximately 36 months.
  DOR: interval from the first documentation of objective tumor regression to the earlier of the first documentation of disease progression or death from any cause.
Progression-free Survival (PFS) | Up to approximately 36 months
  PFS: interval from the start of study drug administration to the earlier of the first documentation of disease progression or death from any cause
Time to Treatment Failure (TTF) | Up to approximately 36 months
  TTF: interval from the start of study drug administration to the earliest of the first documentation of disease progression, the permanent cessation of study drug due to an AE, or death from any cause
Overall Survival (OS) | Up to approximately 36 months
  OS: interval from the start of study drug administration to death from any cause.
SLV-324 Pharmacokinetics: Time to Maximum Concentration (Tmax) | Varying timepoints through the duration of treatment, up to approximately 18 months
  Tmax of SLV-324 antibody-drug conjugate, total antibody, and free payload
SLV-324 Pharmacokinetics: Area Under the Curve (AUC) | Varying timepoints through the duration of treatment, up to approximately 18 months
  AUC of SLV-324 antibody-drug conjugate, total antibody, and free payload
SLV-324 Pharmacokinetics: half-life ( t1/2) | Varying timepoints through the duration of treatment, up to approximately 18 months
  t1/2 of SLV-324 antibody-drug conjugate, total antibody, and free payload

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Washington University, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Generation of a clinical study report (CSR) and publication of results are planned but the sponsor does not currently intend to share individual participant data with other researchers.